CLINICAL TRIAL: NCT02785159
Title: A Phase 2, Multicenter, Double Blinded, Randomized, Vehicle Controlled Study to Compare the Safety and Efficacy of IDP-118 Lotion With Tazorac (Tazarotene) Cream, 0.05% in the Treatment of Plaque Psoriasis
Brief Title: Safety and Efficacy of IDP-118 Lotion in the Treatment of Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: V01-118A-202
Record Dates: First submitted 2016-04-26; First posted 2016-05-27 (Estimated); Results first posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — tazarotene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- IDP-118 Lotion (Experimental): Lotion
  Interventions: Drug: IDP-118 Lotion
- Tazorac Cream (Active Comparator): Cream
  Interventions: Drug: Tazorac Cream
- IDP 118 Vehicle Lotion (Active Comparator): Lotion
  Interventions: Drug: IDP-118 Vehicle Lotion
- IDP-118 Vehicle Cream (Active Comparator): Cream
  Interventions: Drug: IDP-118 Vehicle Cream

INTERVENTIONS:
Drug: IDP-118 Lotion — Lotion
  Other Names: Lotion
  Arms: IDP-118 Lotion
Drug: Tazorac Cream — Cream
  Other Names: Tazorac
  Arms: Tazorac Cream
Drug: IDP-118 Vehicle Lotion — Lotion
  Other Names: Vehicle
  Arms: IDP 118 Vehicle Lotion
Drug: IDP-118 Vehicle Cream — Cream
  Other Names: Vehicle
  Arms: IDP-118 Vehicle Cream

SUMMARY:
Safety and Efficacy of IDP-118 Lotion in the Treatment of Plaque Psoriasis

DETAILED DESCRIPTION:
A Phase 2, Multicenter, Double-Blinded, Randomized, Vehicle-Controlled Study to Compare the Safety and Efficacy of IDP-118 Lotion with Tazorac (tazarotene) Cream, 0.05% in the Treatment of Plaque Psoriasis

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female, of any race, at least 18 years of age (inclusive).
* Freely provides both verbal and written informed consent.
* Has an area of plaque psoriasis appropriate for topical treatment that covers a Body Surface Area (BSA) of at least 3%, but no more than 12%. The face, scalp, palms, soles, axillae, and intertriginous areas are to be excluded in this calculation.
* Is willing and able to avoid prolonged exposure of the treatment area to ultraviolet radiation (natural and artificial) for the duration of the study.
* Has a clinical diagnosis of psoriasis at the Baseline visit with an (IGA) Investigator Global Assessment score of 3 or 4. (The face, scalp, palms, soles, axillae and intertriginous areas are to be excluded in this assessment, if psoriasis is present.)

Key Exclusion Criteria:

* Has spontaneously improving or rapidly deteriorating plaque psoriasis or pustular psoriasis, as determined by the investigator.
* Presents with psoriasis that was treated with prescription medication and failed to respond to treatment, even partially or temporarily, as determined by the investigator.
* Presents with any concurrent skin condition that could interfere with the evaluation of the treatment areas, as determined by the investigator.
* Is pregnant, nursing an infant, or planning a pregnancy during the study period.
* Has received treatment with any investigational drug or device within 60 days or 5 drug half-lives (whichever is longer) prior to the Baseline visit, or is concurrently participating in another clinical study with an investigational drug or device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2016-02; Primary Completion 2016-11-20 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Binu J Alexander, MD, Study Director — Valeant Pharmaceuticals
Locations (14):
- United States (14):
  - Valeant Site 12, Encino, California
  - Valeant Site 13, Orange Park, Florida
  - Valeant Site 11, Pinellas Park, Florida
  - Valeant Site 01, Tampa, Florida
  - Valeant Site 04, Tampa, Florida
  - Valeant Site 05, Plainfield, Indiana
  - Valeant Site 09, Clarkston, Michigan
  - Valeant Site 07, Fridley, Minnesota
  - Valeant Site 14, Saint Joseph, Missouri
  - Valeant Site 10, Greenville, South Carolina
  - Valeant Site 03, Murfreesboro, Tennessee
  - Valeant Site 06, College Station, Texas
  - Valeant Site 08, Webster, Texas
  - Valeant Site 02, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IDP-118 Lotion | Tazorac Cream | IDP 118 Vehicle Lotion | IDP-118 Vehicle Cream
Started | 62 | 58 | 15 | 17
Completed | 51 | 45 | 12 | 14
Not Completed | 11 | 13 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDP-118 Lotion | Tazorac Cream | IDP 118 Vehicle Lotion | IDP-118 Vehicle Cream | Total
Number analyzed (Participants) | 62 | 58 | 15 | 17 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (14.58) | 48.4 (12.37) | 48.9 (14.78) | 56.8 (11.92) | 49.81 (13.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 24 | 7 | 5 | 56
  Male | 42 | 34 | 8 | 12 | 96

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects With Treatment Success, Defined by at Least a 2 Grade Improvement From Baseline in the Investigator Global Assessment (IGA) Score Equating to Clear or Almost Clear.
Description: Treatment success defined as at least a 2-grade improvement from Baseline in the Investigator's Global Assessment (IGA) score and an IGA score equating to "clear" or "almost clear". The IGA score was based on a 5-point scale ranging from 0 to 4 (0=clear, 1=almost clear, 2=mild, 3=moderate, and 4=severe).
Time Frame: 12 Weeks
Measure: Number; unit: percentage of participants
Arm/Group | IDP-118 Lotion | Tazorac Cream | IDP 118 Vehicle Lotion | IDP-118 Vehicle Cream
Number analyzed (Participants) | 62 | 58 | 15 | 17
percentage of participants | 31.66 | 13.77 | 15.90 | 7.96

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Adverse events were collected from participants who were randomized, received at least 1 confirmed dose of study drug, and had at least 1 post-Baseline safety assessment (Safety Population).
Arm/Group | IDP-118 Lotion | Tazorac Cream | IDP 118 Vehicle Lotion | IDP-118 Vehicle Cream
Serious Adverse Events (participants affected / at risk) | 1/60 | 1/57 | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 10/60 | 8/57 | 4/15 | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IDP-118 Lotion (N=60) | Tazorac Cream (N=57) | IDP 118 Vehicle Lotion (N=15) | IDP-118 Vehicle Cream (N=16)
Chest pain (General disorders) | 1 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IDP-118 Lotion (N=60) | Tazorac Cream (N=57) | IDP 118 Vehicle Lotion (N=15) | IDP-118 Vehicle Cream (N=16)
Skin atrophy (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0
Application site pain (General disorders) | 4 | 3 | 2 | 0
Application site pruritis (General disorders) | 2 | 2 | 2 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.